CLINICAL TRIAL: NCT01257230
Title: A Phase III, Randomised, Double Blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety Over 48 Weeks of Orally Inhaled Tiotropium Bromide (2.5 and 5 µg Once Daily ) Delivered by the Respimat® Inhaler in Adolescents (12 to 17 Years Old) With Moderate Persistent Asthma.
Brief Title: Efficacy and Safety of 2 Doses of Tiotropium Via Respimat Compared to Placebo in Adolescents With Moderate Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.444; 2010-021093-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (3):
- placebo (Placebo Comparator): once daily, delivered with Respimat inhaler
  Interventions: Drug: placebo Respimat
- tiotropium low dose (Experimental): once daily, delivered with Respimat inhaler
  Interventions: Drug: tiotropium Respimat low dose
- tiotropium high dose (Experimental): once daily, delivered with Respimat inhaler
  Interventions: Drug: tiotropium Respimat high dose

INTERVENTIONS:
Drug: tiotropium Respimat low dose — IMP
  Arms: tiotropium low dose
Drug: placebo Respimat — placebo representing comparator
  Arms: placebo
Drug: tiotropium Respimat high dose — IMP
  Arms: tiotropium high dose

SUMMARY:
The aim of the study is to evaluate efficacy and safety of a 48-week treatment with two doses of tiotropium bromide compared to placebo in adolescent patients with moderate persistent asthma. Efficacy and safety will be assessed by measuring lung function parameters and evaluating the effects on asthma exacerbations, on Quality of life, on health care resource utilisation an on the number of adverse events.

ELIGIBILITY:
Inclusion criteria:

1. All patients and their parents (or legally accepted caregiver) must sign and date an informed consent consistent with ICH-GCP guidelines and local legislation prior to participation in the trial.
2. Male or female patients between 12 and 17 years of age.
3. All patients must have at least a 3 months history of asthma at the time of enrolment into the trial. The diagnosis of asthma has to be confirmed at visit 1 with a bronchodilator reversibility test.
4. All patients must have been on maintenance treatment with inhaled corticosteroids at a stable medium dose for at least 4 weeks before Visit 1.
5. All patients must be symptomatic (partly controlled) at Visit 1 (screening) and at randomisation defined by an Asthma Control Questionnaire (ACQ) mean score of more than or equal to 1.5.
6. All patients must have a pre-bronchodilator FEV1 more than or equal to 60% and less than or equal to 90% of predicted normal at Visit 1. Variation of absolute FEV1 values of Visit 1 as compared to Visit 2 must be within ± 30%.
7. All patients must have an increase in FEV1 of equal or above 12% and 200 mL after 400 µg salbutamol (albuterol) at Visit 1. If patients in the lower age range (e.g., 12 to 14 year olds) exhibit a very small total lung volume, positive reversibility testing might be based solely on the relative (12%) post-bronchodilator response.
8. All patients should be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment.
9. Patients should be able to use the Respimat® inhaler correctly.
10. Patients must be able to perform all trial related procedures including technically acceptable spirometric manoeuvres.

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. Patients with clinically relevant abnormal screening haematology or blood chemistry
3. Patients with a history of congenital or acquired heart disease, and/or have been hospitalised for cardiac syncope or failure during the past year.
4. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
5. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
6. Patients with lung diseases other than asthma (e.g. Cystic Fibrosis). In case of ex-premature infants, a history of significant bronchopulmonary dysplasia will be regarded as exclusion criterion.
7. Patients with known active tuberculosis.
8. Patients with significant alcohol or drug abuse within the past two years.
9. Patients who have undergone thoracotomy with pulmonary resection.
10. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1).
11. Patients with known hypersensitivity to anticholinergic drugs, Benzalkonium chloride (BAC), Ethylenediaminetetraacetic acis (EDTA) or any other components of the tiotropium inhalation solution.
12. Pregnant or nursing adolescent female patients
13. Sexually active female patients of child-bearing potential not using a highly effective method of birth control.
14. Patients who have taken an investigational drug within 4 weeks prior to Visit 1.
15. Patients who have been treated with long-acting anticholinergics (e.g. tiotropium -Spiriva) within four weeks prior to screening (Visit 1).
16. Patients who are unable to comply with pulmonary medication restrictions prior to randomisation.
17. Patients who have been treated with Anti-IgE treatment (Omalizumab Xolair) within the last 6 months prior to screening.
18. Patients who have been treated with systemic (oral or intravenous) corticosteroids within 4 weeks prior to screening (Visit 1).
19. Patients who have been treated with long-acting theophylline preparations within 2 weeks prior to screening (Visit 1) or during the run-in period
20. Patients who have been treated with other non-approved and according to international guidelines not recommended ¿experimental¿ drugs for routine asthma therapy.
21. Patients with any acute asthma exacerbation or respiratory tract infection in the 4 weeks prior to Visit 1.
22. Patients requiring 10 or more puffs of rescue medication (salbutamol/albuterol) per day on more than 2 consecutive days during the run-in period.
23. Patients who have previously been randomised in this trial or are currently participating in another study.
24. Patients who are being treated with oral beta-blocker medication.
25. Patients with a known narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
26. Patients with renal impairment, as defined by a creatinine clearance less than 50 mL/min/1.73 m2 Body Surface Area as calculated by Schwartz formula.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 398 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (66):
- United States (8):
  - 205.444.01004 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 205.444.01005 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.444.01001 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.444.01014 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.444.01002 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.444.01012 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.444.01013 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 205.444.01003 Boehringer Ingelheim Investigational Site, South Burlington, Vermont
- Chile (3):
  - 205.444.56002 Boehringer Ingelheim Investigational Site, Santiago
  - 205.444.56001 Boehringer Ingelheim Investigational Site, Viña del Mar
  - 205.444.56003 Boehringer Ingelheim Investigational Site, Viña del Mar
- Germany (6):
  - 205.444.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 205.444.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 205.444.49001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.444.49003 Boehringer Ingelheim Investigational Site, Ettenheim
  - 205.444.49006 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.444.49005 Boehringer Ingelheim Investigational Site, Rosenheim
- Hungary (8):
  - 205.444.36007 Boehringer Ingelheim Investigational Site, Ajka
  - 205.444.36005 Boehringer Ingelheim Investigational Site, Budapest
  - 205.444.36008 Boehringer Ingelheim Investigational Site, Budapest
  - 205.444.36006 Boehringer Ingelheim Investigational Site, Kaposvár
  - 205.444.36001 Boehringer Ingelheim Investigational Site, Miskolc
  - 205.444.36002 Boehringer Ingelheim Investigational Site, Mosdós
  - 205.444.36003 Boehringer Ingelheim Investigational Site, Szeged
  - 205.444.36004 Boehringer Ingelheim Investigational Site, Szigetbecse
- Italy (3):
  - 205.444.39001 Boehringer Ingelheim Investigational Site, Ancona
  - 205.444.39003 Boehringer Ingelheim Investigational Site, Bolzano
  - 205.444.39002 Boehringer Ingelheim Investigational Site, Verona
- Latvia (7):
  - 205.444.37101 Boehringer Ingelheim Investigational Site, Baldone
  - 205.444.37107 Boehringer Ingelheim Investigational Site, Balvi
  - 205.444.37102 Boehringer Ingelheim Investigational Site, Ogre
  - 205.444.37105 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.444.37106 Boehringer Ingelheim Investigational Site, Riga
  - 205.444.37103 Boehringer Ingelheim Investigational Site, Talsi
  - 205.444.37104 Boehringer Ingelheim Investigational Site, Tukums
- Mexico (3):
  - 205.444.52002 Boehringer Ingelheim Investigational Site, Guadalajara
  - 205.444.52001 Boehringer Ingelheim Investigational Site, Hermosillo
  - 205.444.52003 Boehringer Ingelheim Investigational Site, Monterrey
- Russia (6):
  - 205.444.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 205.444.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.444.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.444.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.444.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.444.70001 Boehringer Ingelheim Investigational Site, Yaroslavl
- Slovakia (4):
  - 205.444.42104 Boehringer Ingelheim Investigational Site, Košice
  - 205.444.42106 Boehringer Ingelheim Investigational Site, Martin
  - 205.444.42101 Boehringer Ingelheim Investigational Site, Nitra
  - 205.444.42105 Boehringer Ingelheim Investigational Site, Rožňava
- South Korea (4):
  - 205.444.82003 Boehringer Ingelheim Investigational Site, Guri-si
  - 205.444.82006 Boehringer Ingelheim Investigational Site, Incheon
  - 205.444.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 205.444.82004 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 205.444.34007 Boehringer Ingelheim Investigational Site, Esplugues Del Llobregat
  - 205.444.34001 Boehringer Ingelheim Investigational Site, Madrid
  - 205.444.34004 Boehringer Ingelheim Investigational Site, Majadahonda (Madrid)
  - 205.444.34005 Boehringer Ingelheim Investigational Site, Marbella
  - 205.444.34006 Boehringer Ingelheim Investigational Site, Sabdadell
  - 205.444.34008 Boehringer Ingelheim Investigational Site, Valencia
- Ukraine (8):
  - 205.444.38008 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.444.38002 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.444.38005 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.444.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 205.444.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 205.444.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 205.444.38010 Boehringer Ingelheim Investigational Site, Zaporizhya
  - 205.444.38009 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Halpin DMG, Hamelmann EH, Frith PA, Moroni-Zentgraf PM, van Hecke B, Unseld A, Kerstjens HAM, Szefler SJ. Comparative Responses in Lung Function Measurements with Tiotropium in Adolescents and Adults, and Across Asthma Severities: A Post Hoc Analysis. Pulm Ther. 2020 Jun;6(1):131-140. doi: 10.1007/s41030-020-00113-w. Epub 2020 Mar 16. PMID 32180164
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Hamelmann E, Bateman ED, Vogelberg C, Szefler SJ, Vandewalker M, Moroni-Zentgraf P, Avis M, Unseld A, Engel M, Boner AL. Tiotropium add-on therapy in adolescents with moderate asthma: A 1-year randomized controlled trial. J Allergy Clin Immunol. 2016 Aug;138(2):441-450.e8. doi: 10.1016/j.jaci.2016.01.011. Epub 2016 Mar 5. PMID 26960245

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Respimat: Inhalation of placebo solution once daily for 48 weeks, delivered by the Respimat Inhaler
- Tio R2.5: Inhalation of 2.5μg tiotropium bromide solution once daily for 48 weeks, delivered by the Respimat Inhaler
- Tio R5: Inhalation of 5μg tiotropium bromide solution once daily for 48 weeks, delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Started | 138 | 125 | 135
Completed | 132 | 115 | 129
Not Completed | 6 | 10 | 6
Not completed — Not Treated | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Other reason not defined above | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised patients who were dispensed trial medication and received at least one documented dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 138 | 125 | 134 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.7) | 14.2 (1.8) | 14.5 (1.6) | 14.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 44 | 45 | 139
  Male | 88 | 81 | 89 | 258

OUTCOME MEASURES:

1. Primary Outcome: FEV1 peak0-3 Change From Baseline
Description: Change from baseline in peak Forced expiratory volume in 1 second within the first 3 hours post dosing (FEV1 peak0-3) measured at week 24.
  Note, the measured values presented are actually adjusted means.
Time Frame: Baseline and 24 weeks
Population: Full analysis set (FAS) was the same as the treated set which included all randomised patients who were dispensed trial medication and received at least one documents dose of trial medication. Missing data at a visit was imputed by the available data from the patient at that visit, completely missing visits were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 120 | 131
Litres | 0.373 (0.037) | 0.507 (0.040) | 0.547 (0.038)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis; Mean Difference (Final Values) = 0.134, 95% CI 2-sided [0.034 to 0.234], Standard Error of Mean 0.051 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.076 to 0.272], Standard Error of Mean 0.050 — Difference calculated as Tio R5 minus placebo

2. Secondary Outcome: Trough FEV1 Change From Baseline
Description: Change from baseline in Trough (pre-dose) Forced expiratory volume in 1 second (FEV1) measured at week 24.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 24 weeks
Population: Full analysis set. Missing data at a visit was imputed by the available data from the patient at that visit, completely missing visits were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 119 | 131
Litres | 0.283 (0.040) | 0.367 (0.044) | 0.400 (0.041)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1307, Mixed Models Analysis; Mean Difference (Final Values) = 0.084, 95% CI 2-sided [-0.025 to 0.194], Standard Error of Mean 0.056 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.0320, Mixed Models Analysis; Mean Difference (Final Values) = 0.117, 95% CI 2-sided [0.010 to 0.223], Standard Error of Mean 0.054 — Difference calculated as Tio R5 minus placebo

3. Secondary Outcome: FVC peak0-3 Change From Baseline
Description: Change from baseline in Maximum forced vital capacity (FVC) measured within the first 3 h after administration of trial medication (FVC peak0-3h) after 24 weeks of treatment.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 120 | 131
Litres | 0.331 (0.041) | 0.419 (0.045) | 0.403 (0.043)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1231, Mixed Models Analysis; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [-0.024 to 0.200], Standard Error of Mean 0.057 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1950, Mixed Models Analysis; Mean Difference (Final Values) = 0.072, 95% CI 2-sided [-0.037 to 0.182], Standard Error of Mean 0.056 — Difference calculated as Tio R5 minus placebo

4. Secondary Outcome: Trough FVC Change From Baseline
Description: Change from baseline of Trough (pre-dose) forced vital capacity (FVC) measured 10 min before the administration of trial medication after 24 weeks of treatment.
  The measured values presented are actually adjusted means..
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 119 | 131
Litres | 0.281 (0.043) | 0.345 (0.047) | 0.316 (0.045)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2921, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [-0.055 to 0.181], Standard Error of Mean 0.060 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5495, Mixed Models Analysis; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.080 to 0.150], Standard Error of Mean 0.059 — Difference calculated as Tio R5 minus placebo

5. Secondary Outcome: FEV1 AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 h for FEV1 (FEV1 AUC 0-3h) after 24 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 119 | 131
Litres | 0.281 (0.035) | 0.411 (0.038) | 0.463 (0.036)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0079, Mixed Models Analysis; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [0.034 to 0.225], Standard Error of Mean 0.049 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [0.088 to 0.275], Standard Error of Mean 0.048 — Difference calculated as Tio R5 minus placebo

6. Secondary Outcome: FVC AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 h for FVC (FVC AUC0-3h) after 24 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres
Groups:
- Tio R2.5: Inhalation of 2.5μg tiotropium bromide solution once daily for 48 weeks delivered by the Respimat Inhaler
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 119 | 131
Litres | 0.240 (0.039) | 0.330 (0.042) | 0.311 (0.040)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0945, Mixed Models Analysis; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.016 to 0.196], Standard Error of Mean 0.054 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1755, Mixed Models Analysis; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.032 to 0.175], Standard Error of Mean 0.053 — Difference calculated as Tio R5 minus placebo

7. Secondary Outcome: FEF25-75 Change From Baseline
Description: Change from baseline in mean forced expiratory flow between 25% and 75% of the FVC (FEF25-75%), also known as maximum mid-expiratory flow, at individual time points after 24 weeks of treatment.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Litres per second
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 137 | 120 | 131
Litres per second
  10 minutes pre-dose (n=137, 119, 131) | 0.332 (0.072) | 0.461 (0.079) | 0.609 (0.074)
  30 minutes post-dose | 0.372 (0.066) | 0.536 (0.072) | 0.763 (0.068)
  1 hour post-dose | 0.359 (0.067) | 0.596 (0.072) | 0.835 (0.069)
  2 hours post-dose | 0.403 (0.069) | 0.615 (0.075) | 0.857 (0.071)
  3 hours post-dose | 0.347 (0.068) | 0.653 (0.074) | 0.850 (0.070)

8. Secondary Outcome: Use of PRN Rescue Medication During the Daytime
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the daytime based on the weekly mean at week 24.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and Week 24
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 114 | 122
Number of puffs of rescue medication | -0.206 (0.066) | -0.209 (0.071) | -0.215 (0.068)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9760, Mixed Models Analysis; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.184 to 0.178], Standard Error of Mean 0.092 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.9224, Mixed Models Analysis; Mean Difference (Final Values) = -0.009, 95% CI 2-sided [-0.186 to 0.168], Standard Error of Mean 0.090 — Difference calculated as Tio R5 minus placebo

9. Secondary Outcome: Use of PRN Rescue Medication During the Night-time
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the night-time based on the weekly mean at week 24.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and week 24
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 110 | 124
Number of puffs of rescue medication | -0.144 (0.059) | -0.122 (0.064) | -0.032 (0.061)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.7852, Mixed Models Analysis; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.140 to 0.185], Standard Error of Mean 0.083 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1649, Mixed Models Analysis; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [-0.046 to 0.271], Standard Error of Mean 0.081 — Difference calculated as Tio R5 minus placebo

10. Secondary Outcome: Use of PRN Rescue Medication During the Day
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the day (24 hour period) based on the weekly mean at week 24.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and week 24
Population: FAS
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 117 | 125
Number of puffs of rescue medication | -0.524 (0.098) | -0.556 (0.104) | -0.480 (0.100)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8253, Mixed Models Analysis; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.312 to 0.249], Standard Error of Mean 0.143 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7559, Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.232 to 0.319], Standard Error of Mean 0.140 — Difference calculated as Tio R5 minus placebo

11. Secondary Outcome: Control of Asthma as Assessed by ACQ Total Score
Description: Change from baseline in Asthma Control Questionnaire (ACQ) total score measured at week 24.
  The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ total score was calculated as the mean of the responses to all 7 questions.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and week 24
Population: FAS
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 136 | 120 | 132
Units on a scale | 1.213 (0.062) | 1.053 (0.067) | 1.116 (0.064)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0653, Mixed Models Analysis; Mean Difference (Final Values) = -0.160, 95% CI 2-sided [-0.330 to 0.010], Standard Error of Mean 0.087 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2516, Mixed Models Analysis; Mean Difference (Final Values) = -0.097, 95% CI 2-sided [-0.263 to 0.069], Standard Error of Mean 0.084 — Difference calculated as Tio R5 minus placebo

12. Secondary Outcome: ACQ Total Score Responders
Description: Responder rates based on the ACQ total score after 24 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≤-0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≥0.5)
  The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
Time Frame: Week 24
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 138 | 125 | 134
percentage of participants
  Responder | 66.7 | 76.0 | 74.6
  No change | 27.5 | 21.6 | 23.1
  Worsening | 5.8 | 2.4 | 2.2

13. Secondary Outcome: Control of Asthma as Assessed by ACQ6
Description: Change from baseline in AQC6 score at week 24.
  The ACQ6 score is calculated as the mean of the responses to the first 6 questions of the ACQ. The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and week 24
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 136 | 120 | 132
units on a scale | 1.173 (0.068) | 1.026 (0.073) | 1.119 (0.070)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1200, Mixed Models Analysis; Mean Difference (Final Values) = -0.147, 95% CI 2-sided [-0.333 to 0.038], Standard Error of Mean 0.095 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5589, Mixed Models Analysis; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.235 to 0.127], Standard Error of Mean 0.092 — Difference calculated as Tio R5 minus placebo

14. Secondary Outcome: ACQ6 Responders
Description: Responder rates based on the ACQ6 after 24 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≤-0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≥0.5)
  The ACQ6 score is calculated as the mean of the responses to the first 6 questions of the ACQ. The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
Time Frame: Week 24
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 138 | 125 | 134
percentage of participants
  Responder | 69.6 | 76.8 | 72.4
  No change | 22.5 | 20.0 | 23.1
  Worsening | 8.0 | 3.2 | 4.5

15. Secondary Outcome: Time to First Severe Asthma Exacerbation During the 48 Week Treatment Period
Description: The median time to first severe asthma exacerbation was not calculable, so the number of patients who experienced a severe asthma exacerbation are presented for the measured values. A severe asthma exacerbation was defined as a subgroup of all asthma exacerbations that required treatment with systemic corticosteroid for at least 3 days.
Time Frame: 48 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 138 | 125 | 134
Participants | 9 | 5 | 2
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.4023, Regression, Cox; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.21 to 1.87]
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.0620, Regression, Cox; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.05 to 1.08]

16. Secondary Outcome: Time to First Asthma Exacerbation During the 48 Week Treatment Period
Description: The median time to first asthma exacerbation was not calculable, so the number of patients who experienced an asthma exacerbation are presented for the measured values.
Time Frame: Week 48
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 138 | 125 | 134
Participants | 37 | 34 | 30
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8700, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.65 to 1.66]
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.4198, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.51 to 1.33]

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug intake, up to 416 days
Description: Treated set which included all randomised patients who were dispensed trial medication and received at least one documented dose of trial medication.
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 2/138 | 2/125 | 3/134
Other Adverse Events (participants affected / at risk) | 62/138 | 55/125 | 61/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=138) | Tio R2.5 (N=125) | Tio R5 (N=134)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Allergy to plants (Immune system disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=138) | Tio R2.5 (N=125) | Tio R5 (N=134)
Nasopharyngitis (Infections and infestations) | 17 | 13 | 20
Respiratory tract infection viral (Infections and infestations) | 11 | 11 | 10
Tonsillitis (Infections and infestations) | 7 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 7
Viral infection (Infections and infestations) | 6 | 5 | 7
Peak expiratory flow rate decreased (Investigations) | 8 | 9 | 6
Headache (Nervous system disorders) | 2 | 7 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 32 | 27 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.